CLINICAL TRIAL: NCT00398801
Title: Gastroparesis Registry
Acronym: GpR
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: U01DK074008 GpR; U01DK074008 (NIH)
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Gastroparesis
Keywords: gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Gastroparesis Registry (GpR) is an observational study to clarify the epidemiology, natural history, clinical course, and other outcomes of gastroparesis.

DETAILED DESCRIPTION:
The Gastroparesis Registry (GpR) is an observational study to clarify the epidemiology, natural history, clinical course, and other outcomes of gastroparesis. The Gastroparesis Registry will also provide a resource to inform the development of clinical trials and ancillary studies of the epidemiology, etiology, pathophysiology, and impact of gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of gastroparesis of at least 12 weeks duration (do not have to be contiguous) with varying degrees of nausea, vomiting, abdominal pain, early satiety, post-prandial fullness,
* Completion of a 4-hour scintigraphic low fat Egg Beaters gastric emptying study
* Patients with either or both abnormal 2 hour (>60% retention) and 4 hour (>10% retention) gastric emptying will be enrolled and classified as definite gastroparesis (Gp)
* Patients with normal gastric emptying, but with symptoms of gastroparesis may be enrolled and classified as possible gastroparesis or gastroparesis-like with normal gastric emptying (GLNGE)
* Age at least 18 years at initial screening visit
* Ability and willingness to participate in follow-up

Exclusion Criteria:

* Inability to comply with or complete the gastric emptying scintigraphy
* Presence of other conditions that could explain the patient's symptoms:
* Pyloric or intestinal obstruction
* Active inflammatory bowel disease
* Eosinophilic gastroenteritis
* Neurological conditions such as increased intracranial pressure, space occupying or inflammatory/infectious lesions
* Acute liver failure
* Advanced liver disease (Child's B or C)
* Acute renal failure
* Untreated chronic renal failure (serum creatinine >3 mg/dL)
* Total or subtotal gastric resection (patients with prior fundoplication or postvagotomy gastroparesis after pyloroplasty or antrectomy with Billroth I, Billroth II, or Roux-en-Y gastrojejunostomy will be eligible for enrollment)
* Any other plausible structural or metabolic cause
* Any other condition, which in the opinion of the investigator would interfere with study requirements
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care centers for patients with symptoms of gastroparesis
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Tonascia, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; Henry P Parkman, MD, Principal Investigator — Temple University Hospital; William L Hasler, MD, Principal Investigator — University of Michigan; Thomas L Abell, MD, Principal Investigator — University of Mississippi Medical Center; Pankaj J Pasricha, MD, Principal Investigator — Stanford University; Kenneth L Koch, MD, Principal Investigator — Wake Forest University Health Sciences; Richard W McCallum, MD, Principal Investigator — Texas Tech University Health Science Center
Locations (7):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center (TTUHSC), El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/gpr/?query=gpr
Supporting Information: Study Protocol, ICF
Time Frame: Data deposited 05Jul2016
Access Criteria: Registered user of NIDDK Central Repository
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Result] Parkman HP, Yates K, Hasler WL, Nguyen L, Pasricha PJ, Snape WJ, Farrugia G, Koch KL, Calles J, Abell TL, Sarosiek I, McCallum RW, Lee L, Unalp-Arida A, Tonascia J, Hamilton F. Cholecystectomy and clinical presentations of gastroparesis. Dig Dis Sci. 2013 Apr;58(4):1062-73. doi: 10.1007/s10620-013-2596-y. Epub 2013 Mar 2. PMID 23456496
- [Derived] Sarosiek I, Van Natta M, Parkman HP, Abell T, Koch KL, Kuo B, Shulman RJ, Farrugia G, Grover M, Hamilton FA, Pasricha PJ, Yates KP, Miriel L, Wilson L, Yamada G, Tonascia J, McCallum RW; National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Gastroparesis Clinical Research Consortium (GpCRC). Effect of Domperidone Therapy on Gastroparesis Symptoms: Results of a Dynamic Cohort Study by NIDDK Gastroparesis Consortium. Clin Gastroenterol Hepatol. 2022 Mar;20(3):e452-e464. doi: 10.1016/j.cgh.2021.05.063. Epub 2021 Jun 2. PMID 34089855
- [Derived] Pasricha PJ, Grover M, Yates KP, Abell TL, Bernard CE, Koch KL, McCallum RW, Sarosiek I, Kuo B, Bulat R, Chen J, Shulman RJ, Lee L, Tonascia J, Miriel LA, Hamilton F, Farrugia G, Parkman HP; National Institute of Diabetes and Digestive and Kidney Diseases/National Institutes of Health Gastroparesis Clinical Research Consortium. Functional Dyspepsia and Gastroparesis in Tertiary Care are Interchangeable Syndromes With Common Clinical and Pathologic Features. Gastroenterology. 2021 May;160(6):2006-2017. doi: 10.1053/j.gastro.2021.01.230. Epub 2021 Feb 3. PMID 33548234
- [Derived] Parkman HP, Wilson LA, Yates KP, Koch KL, Abell TL, McCallum RW, Sarosiek I, Kuo B, Malik Z, Schey R, Shulman RJ, Grover M, Farrugia G, Miriel L, Tonascia J, Hamilton F, Pasricha PJ; NIDDK/NIH Clinical Gastroparesis Consortium. Factors that contribute to the impairment of quality of life in gastroparesis. Neurogastroenterol Motil. 2021 Aug;33(8):e14087. doi: 10.1111/nmo.14087. Epub 2021 Jan 25. PMID 33493377
- [Derived] Pasricha PJ, Yates KP, Nguyen L, Clarke J, Abell TL, Farrugia G, Hasler WL, Koch KL, Snape WJ, McCallum RW, Sarosiek I, Tonascia J, Miriel LA, Lee L, Hamilton F, Parkman HP. Outcomes and Factors Associated With Reduced Symptoms in Patients With Gastroparesis. Gastroenterology. 2015 Dec;149(7):1762-1774.e4. doi: 10.1053/j.gastro.2015.08.008. Epub 2015 Aug 21. PMID 26299414
- [Derived] Parkman HP, Yates K, Hasler WL, Nguyen L, Pasricha PJ, Snape WJ, Farrugia G, Koch KL, Abell TL, McCallum RW, Lee L, Unalp-Arida A, Tonascia J, Hamilton F; National Institute of Diabetes and Digestive and Kidney Diseases Gastroparesis Clinical Research Consortium. Clinical features of idiopathic gastroparesis vary with sex, body mass, symptom onset, delay in gastric emptying, and gastroparesis severity. Gastroenterology. 2011 Jan;140(1):101-15. doi: 10.1053/j.gastro.2010.10.015. Epub 2010 Oct 20. PMID 20965184
- See also: National Institute of Diabetes and Digestive and Kidney Diseases — http://www2.niddk.nih.gov/
- See also: Gastroparesis Clinical Research Consortium — https://jhuccs1.us/gpcrc/